CLINICAL TRIAL: NCT01232426
Title: A Randomized Controlled Trial of the Treatment of Mallet Fractures: Conservative Versus Operative Using One Meniscus Arrow®
Brief Title: A Randomized Controlled Trial of the Treatment of Mallet Fractures
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Conmed Linvatec Benelux (Other)
Responsible Party: Principal Investigator, Dr. D.B. Wouters, Dr. D.B. Wouters, Conmed Linvatec Benelux
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Mallet2010
Record Dates: First submitted 2010-10-31; First posted 2010-11-02 (Estimated); Last update posted 2012-08-20 (Estimated); Status verified 2012-08

CONDITIONS: Mallet Fracture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Operative (Experimental): operative treatment of a Mallet fracture with a biodegradable Meniscus Arrow®
  Interventions: Procedure: Biodegradable Meniscus Arrow®
- Conservative (Active Comparator): Conservative treatment of a Mallet fracture with a Mallet splint
  Interventions: Device: Mallet splint

INTERVENTIONS:
Procedure: Biodegradable Meniscus Arrow® — Closed reduction of the Mallet fracture and fixation with 1 biodegradable meniscus Arrow®
  Arms: Operative
Device: Mallet splint — Conservative treatment of the Mallet fracture with the traditional Mallet splint.
  Arms: Conservative

SUMMARY:
Intra-articular fractures at the dorsal base of the distal phalanx of the hand are usually referred to as Mallet fractures. Treatment of Mallet fractures remains controversial. Although no differences in clinical results are reported between conservative treatment and operative treatment, operative treatment is suggested for fractures involving more than 30% of articular surface. There are many different operative techniques, all with specific disadvantages. The investigators hypothesis is that operative treatment of Mallet fractures with one Meniscus Arrow® has a better outcome than conservative treatment with a Mallet splint.

ELIGIBILITY:
Inclusion Criteria:

* avulsion fracture involving more than 30% of articular surface

Exclusion Criteria:

* (sub)luxation of the distal phalanx
* patients with a Mallet fracture developed 3 weeks or more prior to presentation
* patients with a Mallet fracture with failure of conservative treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-01 (Estimated)

PRIMARY OUTCOMES:
Extension deficit | 1 year
  To evaluate the extension deficit after conservative and operative treatment of a Mallet fracture using the Crawford criteria.
extension deficit | 1 year
  at every visit, the extension in the DIP joint, is measured

SECONDARY OUTCOMES:
wound healing disturbances | 1 year
  at every control, this is noted

OTHER OUTCOMES:
nail deformaties | 1 year
  at every control nail deformaties, if present, are noted

CONTACTS AND LOCATIONS:
Locations (6):
- Netherlands (6):
  - st. Elisabeth Hospital, Tilburg, Noord-Barbant
  - Amphia Hospital, Breda, North Brabant
  - Catharaina Hospital, Eindhoven, North Brabant
  - Twee Steden Hospital, Tilburg, North Brabant
  - Kennemer Gasthuis Hospital, Haarlem, North Holland
  - Canisius-Wilhelmina Hospital, Nijmegen

REFERENCES:
- [Background] Nelis R, Wouters DB. Is the use of biodegradable devices in the operative treatment of avulsion fractures of fingers, the so-called mallet finger advantageous? A feasibility study with meniscus arrows. Open Orthop J. 2008 Nov 3;2:151-4. doi: 10.2174/1874325000802010151. PMID 19478891